CLINICAL TRIAL: NCT01804309
Title: Functional Anatomical Examination of Axillary Sentinel Lymph Node Drainage in the Axillary Subregions in Early Breast Cancer
Status: Completed | Type: Observational
Sponsor: National Institute of Oncology, Hungary (Other)
Responsible Party: Principal Investigator, Dr. Zoltan Matrai, head of the Dept. of Breast and Sarcoma Surgery, National Institute of Oncology, Hungary
Other Study IDs: FANTON-Ebc
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: axyllary lymph node; sentinel lymph node; lymphatic drainage; early breast cancer; axillary lymph node dissection
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Early breast cancer patients: Clinical stage T1-2 N0M0 primary unilateral invasive breast cancer patients
  Interventions: Procedure: Sentinel lymph node biopsy (SLNB)

INTERVENTIONS:
Procedure: Sentinel lymph node biopsy (SLNB) — The intervention (SLNB) is no different in the care of patients' in the study then in those who were not included in the past or will not be included after the trial terminates. SLNB is performed according to strict professional guidelines adopted by the National Institute of Oncology, Budapest, Hungary.

SUMMARY:
Regional lymph node status is the most important prognostic factor for disease-free and overall survival in breast cancer. Accurate nodal staging can be achieved only by surgery. Today, in early-stage invasive breast cancers with clinically negative lymph nodes, minimally invasive sentinel lymph node biopsy (SLNB) is considered the gold standard of regional lymph node staging. To optimize the effectiveness of SLNB, precise pre-and intraoperative mapping of lymphatic drainage is important. The (SLNB) technique is not standardized. The most common and most accurate way of lymphatic mapping is performed with the combined application of a gamma-emitting isotope labeled substance and blue dye, the so-called double labeling technique. Functional lymphatic drainage of SLNB double staining in the mammary gland, skin and axilla present a number of uncertainties.

According to the axillary, lateral thoracic and thoracodorsal veins, Ibusuki et al. divided the axillary region into four subregions: brachial (lateral), pectoral (anterior), central and subscapular (posterior) zones. They revealed clear relationship between the anatomic location and status of the SLN, also confirmed by Gallowitsch et al. SLN was detected in Level I in 96% and in Level II in 4% by SPECT/CT.

Knowedge of relationships between the drainage of sentinel lymph node staining into the axillary subregions, location of the primary tumor, tumor size, SLN positivity and its location within the subregion are of particular importance in the decision making whether or not axillary lymphadenectomy (ALND) needs to be performed.

In the prospective randomized phase 3 trial by Giuliano et al. (ACOSOG Z-11) ALND was not performed in early breast cancer patients with clinically negative axilla and breast-conserving surgery, for 1-2 macroscopically positive SLNs (10). After an average follow-up of 6.3 years, data were compared to the traditional ALND group and no difference was detected in 5-year overall survival or disease-free survival at 5 years.

Aims of the investigation:

To examine the location of SLN in the axillary subregion (anterior, posterior, central, lateral, apical) in patients with early breast cancer (T <5 cm).

To statistically assess correlations between the location, size, histological parameters of primary breast tumor and the subregion of the SLN.

To statistically assess SLN positivity and its location within the sbregion.

To statistically assess subregional localisation of positive SLN and the number of all positive regional lymph nodes, to predict a limited number of cases with lymph node metastasis, based on the test results of the ACOSOG Z-11 trial, by which ALND could be omitted.

ELIGIBILITY:
Inclusion Criteria:

* women with clinically node negative invasive or microinvasive breast cancer: T1-2(≤ 5cm)N0M0
* 18 years of age or older

Exclusion Criteria:

* previous ALND
* clinically positive axillary SLNB
* pregnant or lactating
* neoadjuvant breast cancer treatment based on surgeon's discretion (ASCO)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical stage T1-2(≤ 5cm)N0M0 primary unilateral invasive breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The assessment of any correlations between the subregional location of SLNs within the axillary trench and the clinical-pathological parameters of the tumor. | Specimen is processed within 2-4 weeks in pathology. Average time frame maximum: 3 weeks following surgical intervention.

SECONDARY OUTCOMES:
The assessment of any correlations between the subregional location of positive SLNs within the axillary trench and the number of all positive axillary lymph nodes. | Same as for primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Zoltán Mátrai, MD, PhD, FEBS, Principal Investigator — National Institute of Oncology; Bence Dorogi, MD, Study Director — National Institute of Oncology
Locations (1):
- National Institute of Oncology, Budapest, Hungary

REFERENCES:
- [Background] Giuliano AE, Haigh PI, Brennan MB, Hansen NM, Kelley MC, Ye W, Glass EC, Turner RR. Prospective observational study of sentinel lymphadenectomy without further axillary dissection in patients with sentinel node-negative breast cancer. J Clin Oncol. 2000 Jul;18(13):2553-9. doi: 10.1200/JCO.2000.18.13.2553. PMID 10893286
- [Background] Matrai Z, Toth L, Saeki T, Sinkovics I, Godeny M, Takeuchi H, Bidlek M, Bartal A, Savolt A, Dorogi B, Kasler M. [The potential role of SPECT/CT in the preoperative detection of sentinel lymph nodes in breast cancer]. Orv Hetil. 2011 Apr 24;152(17):678-88. doi: 10.1556/OH.2011.29077. Hungarian. PMID 21464026
- [Background] Ibusuki M, Yamamoto Y, Kawasoe T, Shiraishi S, Tomiguchi S, Yamashita Y, Honda Y, Iyama K, Iwase H. Potential advantage of preoperative three-dimensional mapping of sentinel nodes in breast cancer by a hybrid single photon emission CT (SPECT)/CT system. Surg Oncol. 2010 Jun;19(2):88-94. doi: 10.1016/j.suronc.2009.04.001. Epub 2009 May 12. PMID 19442515
- [Background] Gallowitsch HJ, Kraschl P, Igerc I, Hussein T, Kresnik E, Mikosch P, Kohlfuerst S, Hausegger K, Lind P. Sentinel node SPECT-CT in breast cancer. Can we expect any additional and clinically relevant information? Nuklearmedizin. 2007;46(6):252-6. PMID 18084680
- [Background] Giuliano AE, Hunt KK, Ballman KV, Beitsch PD, Whitworth PW, Blumencranz PW, Leitch AM, Saha S, McCall LM, Morrow M. Axillary dissection vs no axillary dissection in women with invasive breast cancer and sentinel node metastasis: a randomized clinical trial. JAMA. 2011 Feb 9;305(6):569-75. doi: 10.1001/jama.2011.90. PMID 21304082